CLINICAL TRIAL: NCT01239030
Title: A Randomized, Parallel, Double-Blind Efficacy and Safety Study of Biphentin Methylphenidate HCl Extended Release Capsules Compared to Placebo in Children and Adolescents 6 to 18 Years With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Efficacy and Safety of Methylphenidate HCl ER Capsules in Children and Adolescents With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rhodes Pharmaceuticals, L.P. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RP-BP-EF002
Record Dates: First submitted 2010-11-03; First posted 2010-11-11 (Estimated); Results first posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-01

CONDITIONS: Attention Deficit Hyperactivity Disorder; ADHD
Keywords: inattention; impulsivity; hyperactivity; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Impulsive Behavior; Spasm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 10 mg (Active Comparator): Biphentin Methylphenidate Hydrochloride Extended Release Capsules 10 mg
  Interventions: Drug: Methylphenidate Hydrochloride Extended Release Capsules
- 15 mg (Active Comparator): Biphentin Methylphenidate Hydrochloride Extended Release Capsules 15 mg
  Interventions: Drug: Methylphenidate Hydrochloride Extended Release Capsules
- 20 mg (Active Comparator): Biphentin Methylphenidate Hydrochloride Extended Release Capsules 20 mg
  Interventions: Drug: Methylphenidate Hydrochloride Extended Release Capsules
- 40 mg (Active Comparator): Biphentin Methylphenidate Hydrochloride Extended Release Capsules 40 mg
  Interventions: Drug: Methylphenidate Hydrochloride Extended Release Capsules
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Drug: Placebo
- Methylphenidate HCl ER Capsules (10, 15, 20, 40, 50 or 60 mg) (Experimental): Biphentin Methylphenidate Hydrochloride Extended Release Capsules (10, 15, 20, 40, 50 or 60 mg) - Open Label Phase
  Interventions: Drug: Methylphenidate Hydrochloride Extended Release Capsules

INTERVENTIONS:
Drug: Methylphenidate Hydrochloride Extended Release Capsules — Biphentin Methylphenidate ER Once-A-Day Capsules
  Other Names: Biphentin
  Arms: 10 mg; 15 mg; 20 mg; 40 mg; Methylphenidate HCl ER Capsules (10, 15, 20, 40, 50 or 60 mg)
Drug: Placebo — Placebo capsules
  Other Names: Placebo capsules
  Arms: Placebo

SUMMARY:
This multi-center parallel study is designed to study the efficacy and safety of fixed doses of methylphenidate extended release (ER) capsules of four dose levels compared with a placebo group in pediatric patients with Attention Deficit Hyperactivity Disorder (ADHD) who are between 6 and 18 years old.

DETAILED DESCRIPTION:
This is a parallel, randomized, double-blind, multi-center, placebo-controlled, forced dose, phase 3 study to evaluate the safety and efficacy of Biphentin® methylphenidate hydrochloride (HCl) extended release (ER) capsules in the treatment of Attention Deficit Hyperactivity Disorder (ADHD) in pediatric and adolescent patients aged 6 up to 18 years.

The primary objective was to assess the efficacy of Biphentin compared to placebo, in the clinic setting, as measured by the clinician-administered parent version of the ADHD-RS-IV.

Subjects who met study entry criteria were enrolled in the Double-blind Phase and were randomized to either a fixed dose of Biphentin (!0, 15, 20, or 40 mg/day) or placebo capsule taken daily in the morning for 1 week. Subjects then continued into an Open-label Phase that included dose optimization with doses starting at 10 mg and allowed up to 60 mg. The open-label period following the one double-blind fixed dose week provides additional opportunity for subjects to receive treatment with Biphentin. Extra unscheduled dose optimization visits are allowed as needed for additional dose titration visits during the open-label period.

The safety and tolerability, and efficacy assessments will be conducted throughout the study.

Biphentin® is designed to be a single daily dose alternative to separate doses of immediate release methylphenidate by providing a biphasic plasma profile. It achieves a first Cmax more similar to immediate release methylphenidate.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 6 up to 18
* ADHD diagnosis with ADHD Rating Scale - 4th Edition scores ≥ 90th percentile
* In need of treatment for ADHD and able to have 2-day washout from previous medication
* Females of child-bearing potential not pregnant and practice birth control
* Subject and parent/guardian willing to comply with protocol
* Signed consent and assent

Exclusion Criteria:

* Estimated Full Scale intellectual level below 80 using Wechsler Abbreviated Scale of Intelligence (WASI)
* Current primary psychiatric diagnosis of other listed disorders
* Chronic medical illnesses: seizure, hypertension, thyroid disease, cardiac, family history of sudden death, glaucoma
* Use of psychotropic central nervous system (CNS) meds having effect exceeding 14 days from screening
* Planned use of prohibited drugs
* Is pregnant or breast-feeding
* Significant ECG or laboratory abnormalities
* Experimental drug or medical device within 30 days prior to screening
* Hypersensitivity to methylphenidate
* Inability or unwillingness to comply with protocol
* Well controlled on current ADHD treatment
* Inability to take oral capsules

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 230 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei-wei Chang, Ph.D., Study Director — NuTec Incorporated; Laurence Greenhill, M.D., Principal Investigator — New York State Psychiatric Institute / Columbia University; Sharon B. Wigal, Ph.D., Principal Investigator — University of California, Irvine / Child Development Center; Robert J. Kupper, Ph.D., Study Chair — Rhodes Phamaceuticals, L.P.
Locations (16):
- United States (16):
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - University of California, Irvine/Child Development Center, Irvine, California
  - Synergy Research, National City, California
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Behavioral Clinical Research, Inc., Lauderhill, Florida
  - Martin Kane, DO, Maitland, Florida
  - Segal Institute for clinical Research, North Miami Outpatient Clinic, North Miami, Florida
  - South Shore Psychiatric Services, PC, Marshfield, Massachusetts
  - Precise Research Center, Madison, Mississippi
  - Center for Psychiatry and Behavioural Medicine Inc, Las Vegas, Nevada
  - New York State Psychiatric Institute/Columbia University, New York, New York
  - Department of Psychiatry, Duke University Medical Center, Durham, North Carolina
  - CTMG, New Bern, North Carolina
  - University of Cincinnati College of Medicine/PPSI, Cincinnati, Ohio
  - University Hospital Case Medical Center, Cleveland, Ohio
  - Wharton Research Center, Inc., Wharton, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wigal SB, Nordbrock E, Adjei AL, Childress A, Kupper RJ, Greenhill L. Efficacy of Methylphenidate Hydrochloride Extended-Release Capsules (Aptensio XR) in Children and Adolescents with Attention-Deficit/Hyperactivity Disorder: A Phase III, Randomized, Double-Blind Study. CNS Drugs. 2015 Apr;29(4):331-40. doi: 10.1007/s40263-015-0241-3. PMID 25877989

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 December 2010 (First subject screened) 09 November 2011 (Last subject visit in Open-Label Phase)
Pre-assignment Details: This study planned to randomize approximately 225 subjects to the Double-Blind phase of the study with the goal of approximately 200 subjects completing the double-blind parallel treatment
Groups:
- 10 mg (Double-Blind) Then Methylphenidate HCl ER Capsules 10, 15, 20, 40, 50 or 60 mg (Open Label): Subjects randomized to 10 mg Methylphenidate HCl ER Capsules for 1 week of Double-Blind phase, then entered an 11-week Open Label phase where subject doses were optimized to either Methylphenidate HCl ER Capsules 10, 15, 20, 40, 50 or 60 mg via titration
  Methylphenidate Hydrochloride Extended Release Capsules 10 mg then Methylphenidate Hydrochloride Extended Release Capsules 10, 15, 20, 40, 50 or 60 mg
  Once-A-Day Capsules
- 15 mg (Double-Blind) Then Methylphenidate HCl ER Capsules 10, 15, 20, 40, 50 or 60 mg (Open Label): Subjects randomized to 15 mg Methylphenidate HCl ER Capsules for 1 week of Double-Blind phase, then entered an 11-week Open Label phase where subject doses were optimized to either Methylphenidate HCl ER Capsules 10, 15, 20, 40, 50 or 60 mg via titration
  Methylphenidate Hydrochloride Extended Release Capsules 15 mg then Methylphenidate Hydrochloride Extended Release Capsules 10, 15, 20, 40, 50 or 60 mg
  Once-A-Day Capsules
- 20 mg (Double-Blind) Then Methylphenidate HCl ER Capsules 10, 15, 20, 40, 50 or 60 mg (Open Label): Subjects randomized to 20 mg Methylphenidate HCl ER Capsules for 1 week of Double-Blind phase, then entered an 11-week Open Label phase where subject doses were optimized to either Methylphenidate HCl ER Capsules 10, 15, 20, 40, 50 or 60 mg via titration
  Methylphenidate Hydrochloride Extended Release Capsules 20 mg then Methylphenidate Hydrochloride Extended Release Capsules 10, 15, 20, 40, 50 or 60 mg
  Once-A-Day Capsules
- 40 mg (Double Blind) Then Methylphenidate HCl ER Capsules 10, 15, 20, 40, 50 or 60 mg (Open Label): Subjects randomized to 40 mg Methylphenidate HCl ER Capsules for 1 week of Double-Blind phase, then entered an 11-week Open Label phase where subject doses were optimized to either Methylphenidate HCl ER Capsules 10, 15, 20, 40, 50 or 60 mg via titration
  Methylphenidate Hydrochloride Extended Release Capsules 40 mg then Methylphenidate Hydrochloride Extended Release Capsules 10, 15, 20, 40, 50 or 60 mg
  Once-A-Day Capsules
- Placebo (Double Blind) Then Methylphenidate HCl ER Capsules 10, 15, 20, 40, 50 or 60 mg (Open Label): Subjects randomized Placebo Capsules for 1 week of Double-Blind phase, then entered an 11-week Open Label phase where subject doses were optimized to either Methylphenidate HCl ER Capsules 10, 15, 20, 40, 50 or 60 mg via titration
  Placebo Capsules then Methylphenidate Hydrochloride Extended Release Capsules 10, 15, 20, 40, 50 or 60 mg
  Once-A-Day Capsules
Period: Double Blind
Arm/Group | 10 mg (Double-Blind) Then Methylphenidate HCl ER Capsules 10, 15, 20, 40, 50 or 60 mg (Open Label) | 15 mg (Double-Blind) Then Methylphenidate HCl ER Capsules 10, 15, 20, 40, 50 or 60 mg (Open Label) | 20 mg (Double-Blind) Then Methylphenidate HCl ER Capsules 10, 15, 20, 40, 50 or 60 mg (Open Label) | 40 mg (Double Blind) Then Methylphenidate HCl ER Capsules 10, 15, 20, 40, 50 or 60 mg (Open Label) | Placebo (Double Blind) Then Methylphenidate HCl ER Capsules 10, 15, 20, 40, 50 or 60 mg (Open Label)
Started | 49 | 44 | 45 | 45 | 47
Completed | 48 | 40 | 44 | 43 | 46
Not Completed | 1 | 4 | 1 | 2 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Period: Dose Optimization (Open Label)
Arm/Group | 10 mg (Double-Blind) Then Methylphenidate HCl ER Capsules 10, 15, 20, 40, 50 or 60 mg (Open Label) | 15 mg (Double-Blind) Then Methylphenidate HCl ER Capsules 10, 15, 20, 40, 50 or 60 mg (Open Label) | 20 mg (Double-Blind) Then Methylphenidate HCl ER Capsules 10, 15, 20, 40, 50 or 60 mg (Open Label) | 40 mg (Double Blind) Then Methylphenidate HCl ER Capsules 10, 15, 20, 40, 50 or 60 mg (Open Label) | Placebo (Double Blind) Then Methylphenidate HCl ER Capsules 10, 15, 20, 40, 50 or 60 mg (Open Label)
Started | 48 | 40 | 44 | 43 | 46
Completed | 41 | 38 | 42 | 40 | 39
Not Completed | 7 | 2 | 2 | 3 | 7
Not completed — Adverse Event | 2 | 0 | 2 | 0 | 5
Not completed — Withdrawal by Subject | 4 | 1 | 0 | 2 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 mg | 15 mg | 20 mg | 40 mg | Placebo | Total
Number analyzed (Participants) | 49 | 44 | 45 | 45 | 47 | 230
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 49 | 44 | 45 | 45 | 47 | 230
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.5 (2.89) | 10.2 (3.08) | 11.1 (3.51) | 11.2 (2.49) | 10.9 (3.05) | 10.8 (3.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 14 | 12 | 17 | 76
  Male | 30 | 30 | 31 | 33 | 30 | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 7 | 4 | 3 | 26
  Not Hispanic or Latino | 45 | 36 | 38 | 41 | 44 | 204
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1 | 2
  Asian | 0 | 2 | 0 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 0 | 0 | 2
  Black or African American | 13 | 11 | 9 | 11 | 9 | 53
  White | 34 | 26 | 33 | 32 | 33 | 158
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 3 | 1 | 3 | 12
Region of Enrollment [Number; unit: participants]
  United States | 49 | 44 | 45 | 45 | 47 | 230
ADHD-RS-IV [Mean (Standard Deviation); unit: units on a scale] — Attention Deficit Hyperactivity Disorder Rating Scale-IV (ADHD-RS-IV): The home version of the ADHD-RS-IV comprising symptoms of ADHD was used. This 18-item scale incorporates each of the ADHD symptoms regardless of assigned subtype. Trained clinicians administered questionnaire to parents. Scoring was based on symptom severity on a 4-point scale: 0=never or rarely, 1=sometimes, 2=often, and 3=very often. The Total Score is the sum of the scores for all 18 items, and could range from 0 (no impairment) to 54 (maximal impairment). Lower scores are better outcomes. Population: Baseline analysis is based on efficacy population (N = 221).
  units on a scale
    number analyzed (Participants) | 48 | 40 | 44 | 43 | 46 | 221
    (all) | 37.6 (8.32) | 38.0 (8.64) | 36.2 (8.46) | 35.6 (9.16) | 33.4 (11.01) | 36.1 (9.25)

OUTCOME MEASURES:

1. Primary Outcome: Change in ADHD-RS-IV Total Score From Baseline (Visit 2) to the End of the Double-Blind Phase (Visit 3)
Description: Change in ADHD-RS-IV Total Score from Baseline (Visit 2) to end of Double Blind Phase (Visit 3); [Calculations of baseline values (Visit 2) minus end of Double Blind values (Visit 3), higher differences means better outcomes].
  Attention Deficit Hyperactivity Disorder Rating Scale-IV (ADHD-RS-IV): The home version of the ADHD-RS-IV comprising symptoms of ADHD was used. This 18-item scale incorporates each of the ADHD symptoms regardless of assigned subtype. Trained clinicians administered questionnaire to parents. Scoring was based on symptom severity on a 4-point scale: 0=never or rarely, 1=sometimes, 2=often, and 3=very often. The Total Score is the sum of the scores for all 18 items, and could range from 0 (no impairment) to 54 (maximal impairment).
Time Frame: From baseline (visit 2) to end of of Double-Blind phase (visit 3)
Population: Efficacy Population (N = 221) comprises subjects who completed ADHD-RS-IV assessments on Day 0 and Day 7.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 10 mg: Biphentin Methylphenidate Hydrochloride Extended Release Capsules 10 mg
  Methylphenidate Hydrochloride Extended Release Capsules: Biphentin Methylphenidate ER Once-A-Day Capsules
  Placebo: Placebo Capsules
- 15 mg: Biphentin Methylphenidate Hydrochloride Extended Release Capsules 15 mg
  Methylphenidate Hydrochloride Extended Release Capsules: Biphentin Methylphenidate ER Once-A-Day Capsules
  Placebo: Placebo Capsules
- 20 mg: Biphentin Methylphenidate Hydrochloride Extended Release Capsules 20 mg
  Methylphenidate Hydrochloride Extended Release Capsules: Biphentin Methylphenidate ER Once-A-Day Capsules
  Placebo: Placebo Capsules
- 40 mg: Biphentin Methylphenidate Hydrochloride Extended Release Capsules 40 mg
  Methylphenidate Hydrochloride Extended Release Capsules: Biphentin Methylphenidate ER Once-A-Day Capsules
  Placebo: Placebo Capsules
- Placebo: Placebo capsules
  Methylphenidate Hydrochloride Extended Release Capsules: Biphentin Methylphenidate ER Once-A-Day Capsules
  Placebo: Placebo Capsules
Arm/Group | 10 mg | 15 mg | 20 mg | 40 mg | Placebo
Number analyzed (Participants) | 48 | 40 | 44 | 43 | 46
units on a scale | 9.3 (8.86) | 11.2 (12.06) | 12.3 (9.84) | 13.2 (10.29) | 5.1 (10.29)
Statistical Analysis 1: Comparison: 10 mg vs 15 mg vs 20 mg vs 40 mg vs Placebo; Test type: Superiority or Other; p = 0.0046, ANCOVA

ADVERSE EVENTS:
Time Frame: Treatment-Related Adverse event data during the 12 week study by phase of study. Double Blind phase (one week duration) followed by Open Label phase (11 week duration).
Description: Treatment-Related AEs for Safety Population. Since subjects received multiple dose levels during the open label phase and a subject may have experienced an adverse event which started on one dose level and was ongoing at subsequent dose level(s), the adverse events are presented for all dose levels combined.
Groups:
- Double Blind Phase - Biphentin 10 mg: Double Blind Phase (Week 1) - Biphentin 10 mg: Methylphenidate Hydrochloride Extended Release Capsules 10 mg. Once-A-Day Capsules
- Double Blind Phase - Biphentin 15 mg: Double Blind Phase (Week 1) - Biphentin 15 mg: Methylphenidate Hydrochloride Extended Release Capsules 15 mg. Once-A-Day Capsules
- Double Blind Phase - Biphentin 20 mg: Double Blind Phase (Week 1) - Biphentin 20 mg: Methylphenidate Hydrochloride Extended Release Capsules 20 mg. Once-A-Day Capsules
- Double Blind Phase - Biphentin 40 mg: Double Blind Phase (Week 1) - Biphentin 40 mg: Methylphenidate Hydrochloride Extended Release Capsules 40 mg. Once-A-Day Capsules
- Double Blind Phase - Placebo: Double Blind Phase (Week 1) - Placebo capsules Once daily
- Open Label Phase - Biphentin (10, 15, 20, 30, 40, 50 or 60 mg): Open Label Phase (Week 2-Week 12) - Biphentin Methylphenidate Hydrochloride Extended Release Capsules (10, 15, 20, 30, 40, 50, or 60 mg as directed by Clinician). Once daily
Arm/Group | Double Blind Phase - Biphentin 10 mg | Double Blind Phase - Biphentin 15 mg | Double Blind Phase - Biphentin 20 mg | Double Blind Phase - Biphentin 40 mg | Double Blind Phase - Placebo | Open Label Phase - Biphentin (10, 15, 20, 30, 40, 50 or 60 mg)
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/44 | 0/45 | 0/45 | 0/47 | 0/221
Serious Adverse Events (participants affected / at risk) | 0/49 | 1/44 | 0/45 | 0/45 | 0/47 | 1/221
Other Adverse Events (participants affected / at risk) | 11/49 | 10/44 | 12/45 | 11/45 | 2/47 | 116/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind Phase - Biphentin 10 mg (N=49) | Double Blind Phase - Biphentin 15 mg (N=44) | Double Blind Phase - Biphentin 20 mg (N=45) | Double Blind Phase - Biphentin 40 mg (N=45) | Double Blind Phase - Placebo (N=47) | Open Label Phase - Biphentin (10, 15, 20, 30, 40, 50 or 60 mg) (N=221)
Adjustment disorder with mixed disturbance or emotion and conduct (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Not related to study drug
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 — Not related to study drug - INJURY INDUCED MIGRAINE HEADACHE
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind Phase - Biphentin 10 mg (N=49) | Double Blind Phase - Biphentin 15 mg (N=44) | Double Blind Phase - Biphentin 20 mg (N=45) | Double Blind Phase - Biphentin 40 mg (N=45) | Double Blind Phase - Placebo (N=47) | Open Label Phase - Biphentin (10, 15, 20, 30, 40, 50 or 60 mg) (N=221)
headache (Nervous system disorders) | 5 | 3 | 6 | 5 | 1 | 31
Insomnia (Nervous system disorders) | 4 | 2 | 6 | 5 | 1 | 26
abdominal pain upper (Gastrointestinal disorders) | 3 | 4 | 4 | 1 | 0 | 21
decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 4 | 2 | 0 | 42
fatigue (General disorders) | 2 | 0 | 0 | 0 | 1 | 10
irritability (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 11
Affect Liability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is restricted from using, disclosing, presenting, or publishing trial information without the prior written consent from the Sponsor